CLINICAL TRIAL: NCT00744042
Title: A Multicenter, Open-Label Study of the Safety, Tolerability and Pharmacology of Asfotase Alfa in up to 10 Severely Affected Patients With for the Treatment of Severely Affected Patients With Infantile Hypophosphatasia (HPP)
Brief Title: Safety and Efficacy Study of Asfotase Alfa in Severely Affected Infants With Hypophosphatasia (HPP)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENB-002-08
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Results first posted 2011-09-30 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Hypophosphatasia (HPP)
Keywords: Hypophosphatasia; HPP; Bone Disease; Soft Bones; Low Alkaline Phosphatase; genetic metabolic disorder; alkaline phosphatase; tissue non-specific alkaline phosphatase; rickets; osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- asfotase alfa (Other): asfotase alfa
  Interventions: Biological: asfotase alfa

INTERVENTIONS:
Biological: asfotase alfa
  Other Names: Asfotase Alfa was formerly referred to as ENB-0040; Human Recombinant Tissue Nonspecific Alkaline Phosphatase Fusion Protein

SUMMARY:
This clinical trial studies the safety and efficacy of asfotase alfa in infants and young children with infantile onset HPP.

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is a life-threatening, genetic, and ultra-rare metabolic disease characterized by defective bone mineralization and impaired phosphate and calcium regulation that can lead to progressive damage to multiple vital organs, including destruction and deformity of bones, profound muscle weakness, seizures, impaired renal function, and respiratory failure. There are no approved disease-modifying treatments for patients with this disease. There is also limited data available on the natural course of this disease over time, particularly in patients with the juvenile-onset form.

ELIGIBILITY:
Inclusion Criteria:

* Legal guardian(s) must provide informed consent prior to any study procedures
* Documented diagnosis of severe HPP as indicated by:

  * Total serum alkaline phosphatase at least 3 standard deviations (SD) below the mean for age
  * Plasma pyridoxal 5'-phosphate (PLP) at least 4 times the upper limit of normal
  * Radiographic evidence of HPP (hypophosphatasia), characterized by:

    * Flared and frayed metaphyses
    * Severe, generalized osteopenia
    * Widened growth plates
  * One or more HPP-related findings:

    * History or presence of:

      * Non-traumatic post-natal fracture
      * Delayed fracture healing
    * History of elevated serum calcium
    * Functional craniosynostosis with decreased head circumference growth
    * Nephrocalcinosis
    * Respiratory compromise
  * Rachitic chest deformity and/or vitamin B6 dependent seizures
  * Failure to thrive
* Onset of symptoms prior to 6 months of age
* Age ≤ 36 months
* Otherwise medically stable (patient may be on ventilatory support)
* Legal guardian(s) must be willing to comply with the study

Exclusion Criteria:

* History of sensitivity to any of the constituents of the study drug
* Current or prior clinically significant cardiovascular, endocrinologic, hematologic, hepatic, immunologic, metabolic, infectious, urologic, pulmonary, neurologic, dermatologic, renal condition and/or other major disease which, in the opinion of the investigator, precludes study participation
* Treatment with an investigational drug within 1 month prior to the start of study drug administration
* Current enrollment in any other study involving an investigational new drug, device or treatment for HPP (e.g., bone marrow transplantation)
* Low serum calcium, phosphate or 25(OH) vitamin D
* Current evidence of a treatable form of rickets
* Prior treatment with bisphosphonate

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - St. John's Hospital, Springfield, Missouri
  - University of Nebraska Medical Center, Munroe-Meyer Institute, Omaha, Nebraska
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - St. Vincent Hospital, Green Bay, Wisconsin
- The University of Manitoba Health Sciences Centre, Winnipeg, Manitoba, Canada
- Tawam-John Hopkins Hospital, Al Ain City, Abu Dhabi Emirate, United Arab Emirates
- United Kingdom (2):
  - Sheffield Children's Hospital, Sheffield, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland

REFERENCES:
- [Background] Millan JL, Narisawa S, Lemire I, Loisel TP, Boileau G, Leonard P, Gramatikova S, Terkeltaub R, Camacho NP, McKee MD, Crine P, Whyte MP. Enzyme replacement therapy for murine hypophosphatasia. J Bone Miner Res. 2008 Jun;23(6):777-87. doi: 10.1359/jbmr.071213. PMID 18086009
- [Background] Drake MT, Khosla S. Bone-targeted replacement therapy for hypophosphatasia. J Bone Miner Res. 2008 Jun;23(6):775-6. doi: 10.1359/jbmr.080305. No abstract available. PMID 18318644
- [Derived] Padidela R, Yates R, Benscoter D, McPhail G, Chan E, Nichani J, Mughal MZ, Myer C 4th, Narayan O, Nissenbaum C, Wilkinson S, Zhou S, Saal HM. Characterization of tracheobronchomalacia in infants with hypophosphatasia. Orphanet J Rare Dis. 2020 Aug 6;15(1):204. doi: 10.1186/s13023-020-01483-9. PMID 32762706
- [Derived] Whyte MP, Rockman-Greenberg C, Ozono K, Riese R, Moseley S, Melian A, Thompson DD, Bishop N, Hofmann C. Asfotase Alfa Treatment Improves Survival for Perinatal and Infantile Hypophosphatasia. J Clin Endocrinol Metab. 2016 Jan;101(1):334-42. doi: 10.1210/jc.2015-3462. Epub 2015 Nov 3. PMID 26529632
- [Derived] Whyte MP, Greenberg CR, Salman NJ, Bober MB, McAlister WH, Wenkert D, Van Sickle BJ, Simmons JH, Edgar TS, Bauer ML, Hamdan MA, Bishop N, Lutz RE, McGinn M, Craig S, Moore JN, Taylor JW, Cleveland RH, Cranley WR, Lim R, Thacher TD, Mayhew JE, Downs M, Millan JL, Skrinar AM, Crine P, Landy H. Enzyme-replacement therapy in life-threatening hypophosphatasia. N Engl J Med. 2012 Mar 8;366(10):904-13. doi: 10.1056/NEJMoa1106173. PMID 22397652
- See also: Hypophosphatasia Website — http://www.hypophosphatasia.com
- See also: Hypophosphatasia Website for Healthcare Providers — http://www.hypophosphatasia.com/hcp/
- See also: HPP support group — http://www.magicfoundation.org
- See also: US Hypophosphatasia Group (Soft Bones) — http://www.softbones.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was posted on clinicaltrials.gov. Physicians managing the care of infants and young children with a confirmed diagnosis of HPP contacted existing sites or requested assistance with site set up from the sponsor.
Pre-assignment Details: All screened patients met eligibility criteria and were enrolled in the study.
Groups:
- Asfotase Alfa: All patients received an initial single intravenous (IV) infusion of 2 mg/kg asfotase alfa for the first week followed by regular administration of subcutaneous (SC) injections of 1 mg/kg asfotase alfa 3 times/week (total 3 mg/kg/week).
Period: Overall Study
Arm/Group | Asfotase Alfa
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Asfotase Alfa: All enrolled patients receive a single IV (intravenous) dose of Asfotase Alfa of 2 mg/kg followed by 7 days of observation. Following an assessment of safety data by an independent Data Safety Monitoring Board (DSMB), patients begin thrice weekly SC (subcutaneous) injections of Asfotase Alfa at a dose of 1 mg/kg for the remaining 23 weeks of the study.
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.11 (1.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: participants]
  Canada | 1
  United States | 7
  United Arab Emirates | 1
  United Kingdom | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Rickets Severity From Baseline to Week 24, Based on Assessment of Skeletal Radiographs Using Radiologic Global Impression of Change (RGI-C)
Description: A 7-point RGI-C (Radiographic Global Impression of Change) score was used to rate change in rickets severity. Scores ranged from -3 (severe worsening of rickets) to +3 (complete healing of rickets). Only those patients with a minimum score of +2 indicating substantial healing of rickets) were considered "responders". Three pediatric radiologists not affiliated with the conduct of the study performed the ratings. Average scores were derived for each patient at each assessment.
Time Frame: 24 weeks
Population: ITT (intention to treat)
Measure: Median (Full Range); unit: Units on a scale
Groups:
- Asfotase Alfa: All HPP affected infants will receive a single IV (intravenous) dose of Asfotase Alfa of 2 mg/kg followed by 7 days of observation. Following an assessment of safety data by an independent Data Safety Monitoring Board (DSMB), patients will then begin every other day SC (subcutaneous) injections of Asfotase Alfa at a dose of 1 mg/kg for 23 weeks. End of Study will be at 24 weeks.
Arm/Group | Asfotase Alfa
Number analyzed (Participants) | 11
Units on a scale | 2.00 [0.00 to 2.33]
Statistical Analysis 1: Comparison: Asfotase Alfa; One treatment group; Test type: Superiority or Other; p = 0.0039, Wilcoxon signed-rank test — Testing whether median change in rickets severity from Baseline to Week 24, measured by RGI-C at Week 24, is from zero; The last post-baseline observation carry forward method is used; patients with no post-baseline assessments were imputed as having no change

2. Secondary Outcome: Maximum Serum Concentration of Asfotase Alfa (Cmax)
Description: Maximum serum concentration observed during intensive PK sampling interval.
Time Frame: Study Week 1 (0 to 168 hours post-dose). Study Week 2 and Study Week 3 (0 to 48 hours post-dose)
Population: ITT population. N=number of patients who received a full dose of asfotase alfa and had sufficient data for non-compartmental analysis.
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Study Week 1 Intravenous Dose (2 mg/kg Single Dose): Participants received intravenous (IV) asfotase alfa (2 mg/kg single dose) on Day 1. PK samples drawn predose to 168 hours post-dose.
- Study Week 2 Subcutaneous Dose (1 mg/kg 3x/Week): Participants received subcutaneous (SC) asfotase alfa starting on Day 8 (Week 2) (1 mg/kg 3x/week). PK samples drawn predose to 48 hours post-dose for PK analysis following single SC dose.
- Study Week 3 Subcutaneous Dose (1 mg/kg 3x/Week): Participants received subcutaneous (SC) asfotase alfa starting on Day 8 (Week 2) (1 mg/kg 3x/week). PK samples drawn predose to 48 hours post-dose for PK analysis following multiple SC doses.
Arm/Group | Study Week 1 Intravenous Dose (2 mg/kg Single Dose) | Study Week 2 Subcutaneous Dose (1 mg/kg 3x/Week) | Study Week 3 Subcutaneous Dose (1 mg/kg 3x/Week)
Number analyzed (Participants) | 6 | 7 | 7
U/L | 2230 (1100) | 376 (226) | 897 (491)

3. Secondary Outcome: Time at Maximum Serum Concentration of Asfotase Alfa (Tmax)
Description: Time at maximum serum concentration observed during intensive PK sampling interval.
Time Frame: Study Week 1 (0 to 168 hours post-dose). Study Week 2 and Study Week 3 (0 to 48 hours post-dose).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Groups:
- Study Week 3 Subcutaneous Dose (1mg/kg 3x/Week): Participants received subcutaneous (SC) asfotase alfa starting on Day 8 (Week 2) (1 mg/kg 3x/week). PK samples drawn predose to 48 hours post-dose for PK analysis following multiple SC doses.
Arm/Group | Study Week 1 Intravenous Dose (2 mg/kg Single Dose) | Study Week 2 Subcutaneous Dose (1 mg/kg 3x/Week) | Study Week 3 Subcutaneous Dose (1mg/kg 3x/Week)
Number analyzed (Participants) | 6 | 7 | 7
hour | 4.3 (4.3) | 29.7 (13.2) | 12.0 (7.7)

4. Secondary Outcome: Area Under Serum Concentration-time Curve to Last Measurable Concentration of Asfotase Alfa (AUCt)
Description: Area under serum concentration-time curve to last measurable concentration during intensive PK sampling interval.
Time Frame: Study Week 1 (0 to 168 hours post-dose). Study Week 2 and Study Week 3 (0 to 48 hours post-dose).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*U/L
Groups:
- Study Week 1 Intravenous Dose (2mg/kg Single Dose): Participants received intravenous (IV) asfotase alfa (2mg/mg single dose) on Day 1. PK samples drawn predose to 168 hours post-dose.
- Study Week 2 Subcutaneous Dose (1mg/kg 3x/Week): Participants received subcutaneous (SC) asfotase alfa starting on Day 8 (Week 2) (1 mg/kg 3x/week). PK samples drawn predose to 48 hours post-dose for PK analysis following single SC dose.
Arm/Group | Study Week 1 Intravenous Dose (2mg/kg Single Dose) | Study Week 2 Subcutaneous Dose (1mg/kg 3x/Week) | Study Week 3 Subcutaneous Dose (1mg/kg 3x/Week)
Number analyzed (Participants) | 6 | 7 | 7
h*U/L | 79800 (21700) | 14700 (9730) | 33700 (19700)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Asfotase Alfa: All patients who received any asfotase alfa treatment, regardless of whether they were lost to follow-up or dropped out of the trial.
Arm/Group | Asfotase Alfa
Serious Adverse Events (participants affected / at risk) | 7/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asfotase Alfa (N=11)
H1N1 Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3)
Gastroenteritis salmonella (Infections and infestations) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Craniosynostosis (Congenital, familial and genetic disorders) | 3 (3)
Collapse of lung (Injury, poisoning and procedural complications) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Medical device complication (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asfotase Alfa (N=11)
Pyrexia (General disorders) | 5 (5)
Irritability (General disorders) | 4 (4)
Injection site erythema (General disorders) | 2 (15)
Catheter site erythema (General disorders) | 1 (1)
Catheter site rash (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Injection site hematoma (General disorders) | 1 (4)
Injection site induration (General disorders) | 1 (2)
Injection site nodule (General disorders) | 1 (2)
Injection site pain (General disorders) | 1 (1)
Injection site papule (General disorders) | 1 (1)
Injection site pruritis (General disorders) | 1 (2)
Injection site rash (General disorders) | 1 (2)
Injection site warmth (General disorders) | 1 (2)
Edema (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (4)
Otitis media (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (4)
Bacterial tracheitis (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (2)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Skin candida (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival erythema (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Teething (Gastrointestinal disorders) | 1 (1)
Hemoglobin decreased (Investigations) | 4 (9)
Urine calcium/creatinine ratio increased (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Bradycardia (Cardiac disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Food intolerance (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Drug dependence (Psychiatric disorders) | 3 (3)
Agitation (Psychiatric disorders) | 2 (2)
Breath holding (Psychiatric disorders) | 1 (1)
Congenital bowing of long bones (Congenital, familial and genetic disorders) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 (6)
Piloerection (Skin and subcutaneous tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Ocular hyperaemia (Eye disorders) | 1 (1)
Central venous catheter removal (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Craniosynostosis (Congenital, familial and genetic disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1)
Culture positive (Investigations) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Metabolis acidosis (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Secondary hypertension (Vascular disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less